CLINICAL TRIAL: NCT02158949
Title: Mobilizing to Reduce Overuse of Alcohol in Emergency Department Patients
Brief Title: Study of Mobile Phone Delivered Intervention to Reduce Alcohol Consumption
Acronym: mROAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Burner, Assistant Professor of Clinical Emergency Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-14-00335
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Abuse
Keywords: alcohol; mHealth; SBIRT
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mROAD (Experimental): 1 week of twice daily text messages modeled after SBIRT interventions
  Interventions: Behavioral: mROAD
- Usual Care (No Intervention): Usual care in ED

INTERVENTIONS:
Behavioral: mROAD
  Arms: mROAD

SUMMARY:
In this study, the investigators will be developing and testing a mobile phone text message intervention to reduce alcohol use for people at risk of alcohol dependence. The investigators hypothesize that this intervention will be acceptable to participants, and that they will stay in the intervention until it's one week completion.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT score 15-20
* have a mobile phone capable of receiving text messages

Exclusion Criteria:

* age <18
* unable to consent
* language other than English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05-01; Primary Completion 2014-07-15 (Actual); Study Completion 2014-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Burner, MD MPH, Principal Investigator — University of Southern California
Locations (1):
- LAC+USC Medicine Center Emergency Department, Los Angeles, California, United States

REFERENCES:
- [Derived] Burner E, Zhang M, Terp S, Ford Bench K, Lee J, Lam CN, Torres JR, Menchine M, Arora S. Feasibility and Acceptability of a Text Message-Based Intervention to Reduce Overuse of Alcohol in Emergency Department Patients: Controlled Proof-of-Concept Trial. JMIR Mhealth Uhealth. 2020 Jun 4;8(6):e17557. doi: 10.2196/17557. PMID 32496203

RESULTS

PARTICIPANT FLOW:
Groups:
- mROAD: 1 week of twice daily text messages modeled after SBIRT interventions
  mROAD
Period: Overall Study
Arm/Group | mROAD | Usual Care
Started | 24 | 24
Completed | 18 | 13
Not Completed | 6 | 11
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mROAD | Usual Care | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (13.5) | 35.4 (10.6) | 37.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 19 | 21 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 21 | 38
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 17 | 22 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Self report of mental illness [Count of Participants; unit: Participants] | 6 | 3 | 9
Days drank alcohol in last month [Mean (Standard Deviation); unit: days] | 7.6 (8.6) | 11.5 (8.4) | 9.6 (8.6)
Days drank heavily in last month [Mean (Standard Deviation); unit: days] | 4.9 (7.2) | 5.5 (7.1) | 5.2 (7.1)
Motivation to change score [Mean (Standard Deviation); unit: units on a scale] — Participants reported desire to change via the Change Questionnaire applied to risky alcohol use.[1] The Change questionnaire has a Cronbach's alpha of 0.86 when applied to alcohol use.[2] Minimum score is 0 (low motivation to change) to maximum 120 (high motivation to change).
  1. Miller WR, Johnson WR. A natural language screening measure for motivation to change. Addictive behaviors. 2008;33(9):1177-1182.
  2. Miller WR, Johnson WR. A natural language screening measure for motivation to change. Addictive Behaviors. 2008;33(9):1177-1182.
  units on a scale | 88.8 (6.7) | 89.3 (33.8) | 89.1 (32.9)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention to Patient
Description: percentage of patients that do not opt out of messages prior to 1 week completion
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | mROAD | Usual Care
Number analyzed (Participants) | 24 | 24
Participants | 23 | 24

2. Secondary Outcome: Number of Participants Completed Assessment at 1 Month
Description: Feasibility of follow up of urban low-income at risk drinkers by phone defined as number of patients can be contacted at one months to complete assessment of alcohol use
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | mROAD | Usual Care
Number analyzed (Participants) | 24 | 24
Participants | 18 | 13

3. Secondary Outcome: Change in Days Drinking Alcohol
Description: patients reported number of days drinking any alcohol in prior 30 days, baseline report minus 1 month follow up report
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | mROAD | Usual Care
Number analyzed (Participants) | 18 | 13
days | 2.5 [-1.7 to 6.7] | 8.5 [3 to 13.9]

4. Secondary Outcome: Change in Days Drinking Heavily in 30 Days
Description: patients reported number of heavy drinking days in prior 30 days (3 or more standard sized drinks per episode for women and 4 or more standard sized drinks per episode for men), baseline report minus 1 month follow up report
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | mROAD | Usual Care
Number analyzed (Participants) | 18 | 13
days | 3 [-.7 to 6.7] | 5.6 [-.1 to 11.4]

5. Secondary Outcome: Change in Motivation to Change Score
Description: Participants reported desire to change via the Change Questionnaire applied to risky alcohol use.[1] The Change questionnaire has a Cronbach's alpha of 0.86 when applied to alcohol use.[2] Minimum score is 0 (low motivation to change) to maximum 120 (high motivation to change).
  1. Miller WR, Johnson WR. A natural language screening measure for motivation to change. Addictive behaviors. 2008;33(9):1177-1182.
  2. Miller WR, Johnson WR. A natural language screening measure for motivation to change. Addictive Behaviors. 2008;33(9):1177-1182.
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | mROAD | Usual Care
Number analyzed (Participants) | 18 | 13
score on a scale | 7.6 [-1.7 to 17] | 16.6 [-1.6 to 34]

ADVERSE EVENTS:
Arm/Group | mROAD | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
This is a small pilot trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No